CLINICAL TRIAL: NCT07220629
Title: A Phase 2a Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Explore the Safety and Efficacy of NT-0796 as an Adjunct to Semaglutide Plus a Reduced Calorie Diet and Increased Physical Activity in Participants With Obesity
Brief Title: Study to Explore the Safety and Efficacy of NT-0796 as an Adjunct to Semaglutide in Participants With Obesity (RESOLVE-2)
Acronym: RESOLVE-2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NodThera Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NT-0796-P006
Record Dates: First submitted 2025-10-17; First posted 2025-10-24 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Obesity
Keywords: RESOLVE -2; Obesity; NLRP3; NT-0796
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Twice daily orally administered NT-0796 capsule (Experimental): Participants will receive study medication twice daily orally for up to 20 weeks, containing NT-0796 twice daily
  Interventions: Drug: NT-0796
- Placebo orally administered capsule (Placebo Comparator): Participants will receive placebo twice daily orally for up to 20 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NT-0796 — Orally administered capsules
  Arms: Twice daily orally administered NT-0796 capsule
Drug: Placebo — Orally administered capsules
  Arms: Placebo orally administered capsule

SUMMARY:
A Phase 2a randomized, double-blind, placebo-controlled, parallel-group, multicenter study to explore the safety and efficacy of NT-0796 as an adjunct to semaglutide in participants with obesity over a 6 months treatment period.

DETAILED DESCRIPTION:
Potential participants will be screened within 28 days prior to baseline (Day 1), and eligible participants will be randomly assigned to receive the Investigational Medicinal Product (IMP, either NT-0796 or placebo) twice daily (BID). All participants will receive sc semaglutide. The IMP will be administered orally. Semaglutide will be initiated and titrated using a fixed, 4-weekly dose escalation scheme, as per the approved USPI.

Following 20 weeks of active treatment, participants will enter a 4-week safety follow-up period before being discharged from the study. Semaglutide will be provided for the period from baseline (Day 1) up until completion of the 4-week safety follow-up.

The Primary Endpoint of the study will be the safety and tolerability of NT-0796 as an adjunct to semaglutide, the key secondary endpoint will be the effect of NT-0796 as an adjunct to semaglutide on weight loss while secondary endpoints include percentage weight change from baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 75 years (inclusive) at Screening who have signed informed consent and are willing and able to comply with the study protocol.
2. Have a BMI of ≥30.0 kg/m2 and <45.0 kg/m2 at Screening. (BMI values should be calculated to one decimal point precision and then assessed in terms of the required range).
3. History of at least one self-reported unsuccessful dietary effort to lose body weight.
4. Meeting requirements for, and intending to start, treatment with sc semaglutide, as per the approved USPI.

Exclusion Criteria:

1. Exposure to incretins, irrespective of the indication, within the 12 months prior to Screening.
2. Known hypersensitivity to semaglutide or any of its excipients, or previous inability to tolerate semaglutide.
3. Type 1 or Type 2 Diabetes Mellitus (T1DM or T2DM), and/or HbA1c ≥6.5% (48 mmol/mol) at Screening and/or use of any anti-diabetic medications.
4. History of stroke with residual neurological deficit within 2 years or transient ischemic attack within 6 months prior to Day 1.
5. History of acute coronary syndrome (ACS) including unstable angina, acute myocardial infarction (both ST segment elevation and non-ST segment elevation) within 6 months prior to Day 1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Assess the safety and tolerability of NT-0796 as an adjunct to semaglutide in participants with obesity by assessing AEs and SAEs, symptoms of nausea and vomiting, clinical laboratory parameters, vital signs and ECGs. | Baseline to Week 24

SECONDARY OUTCOMES:
Percent change in body weight in participants with obesity | Baseline to Week 20
Percent change in body weight in participants with obesity | Baseline to Weeks 4, 8, 12, 16, and 24
Change in waist circumference and waist/height ratio | Baseline to Weeks 4, 8, 12, 16, 20, and 24
Proportion of participants that achieve a body weight reduction of ≥5%, ≥10% or ≥15% | Baseline to Week 20
NT-0796/NDT-19795 concentrations in plasma | Baseline to Week 24

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Investigative Site, Mesa, Arizona
  - Investigative Site, Cooper City, Florida
  - Investigative Site, Hialeah, Florida
  - Investigative Site, Jacksonville, Florida
  - Investigative Site, Miami, Florida
  - Investigative Site, Marrero, Louisiana
  - Investigative Site, Columbus, Ohio
  - Investigative Site, Seabrook, Texas
  - Investigative Site, Salt Lake City, Utah
  - Investigative Site, Manassas, Virginia